CLINICAL TRIAL: NCT04715269
Title: Effect of Alprazolam on Heart Rate and Acute Inflammatory Marker in Acute Coronary Syndrome Patients
Brief Title: Role of Alprazolam in the Management of Acute Coronary Syndrome
Acronym: A-ACS-PK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Registrar Cardiology, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZMC/IRB/0022
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Heart Diseases; Anxiety
Keywords: Cardiology; Acute Coronary Syndrome; Heart Rate; Alprazolam; Anxiolytic
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Heart Diseases; Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: This randomized, close label, placebo-controlled study with superiority framework as add-on therapy in ACS patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be done for all participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alprazolam Arm (Experimental): 0.5mg Alprazolam will be given to the patient at the time of presentation
  Interventions: Drug: Alprazolam
- Placebo Arm (Placebo Comparator): The empty capsule will be given to the patient at the time of presentation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprazolam — Alprazolam 0.5 mg will be given when the patient with acute coronary syndrome would present to the emergency
  Arms: Alprazolam Arm
Other: Placebo — Empty capsule
  Arms: Placebo Arm

SUMMARY:
Cardiovascular disease has always been one of the most concerning ailments of all times considering mortality. On one end due to the emergence of pharmaceutical technology, there is a reduction in mortality, on the other hand owing to a sedentary lifestyle the incidence of this disease is increasing. Hence leading to up slopping trend in cardiovascular prevalence. Acute coronary syndrome is one of the most deadly and acute presentations of cardiology requiring immediate intervention to dampen the frequency of complications. One of the fundamental goals in the treatment of ACS is to lower the heart rate so that load on myocardial tissue can be reduced. In order to do so, we already have multiple options like beta-blockers, calcium channel blockers, and new generation ivabradine (not affecting blood pressure unlike others).

DETAILED DESCRIPTION:
World has studied the increased prevalence of anxiety as a concomitant factor in ACS patients causing detrimental effects on cardiovascular outcomes being anxiety as one of the first responses to chest pain and hospital admission causing tachycardia. This study is designed to achieve the goals of lowering the heart using the anxiolytic property of alprazolam. This randomized, parallel group, close label, placebo-controlled, event driven, interventional clinical superiority study will be conducted in Cardiology department of Shaikh Zayed Hospital with a sample size of 48 allocating using lottery method in both experimental and control group. Heart Rate at baseline and after 6 hours will be monitored in both groups to establish the fall of heart rate in both patients. Data will be collected by using pre-designed performa and will be entered and analyzed via SAS 9.4. Statistical analysis will be done using T-test and p value <0.05 will be considered significant.

Significance of the study is to lower the required dosage of beta-blockers in order to achieve optimum beta-blockade using an anxiolytic while not affecting the blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Systolic BP>100mm Hg Age between 18-80 years Sinus Rhythm

Exclusion Criteria:

* Cardiogenic Shock / Hypotension
* Known Asthma/COPD
* Bradycardia (HR < 60)
* Already on Beta blockers/ Anxiolytics
* Sick sinus syndrome
* Second or third-degree heart block (in the absence of pacemaker)
* Decompensated heart failure
* With documented hypersensitivity to the drug or components
* Valvular Heart Diseases
* Congenital Heart Diseases
* Status post CABG
* Any co-morbidities except Diabetes Mellitus and Hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | upto 72 hours
  Heart Rate reduction
Duration of Hospital stay | upto 14 days
  Number of days
Mortality | upto 14 days
  death of patients
recurrent symptomatic ischemia | 72 hours
  episodes of angina
erythrocyte sedimentation rate (ESR) | upto 72 hours
  Acute phase reactants
C-reactive protein (CRP) | upto 72 hours
  Acute phase reactants

CONTACTS AND LOCATIONS:
Overall Officials: Qazi Abdul Saboor, MBBS, Study Chair — Shaikh Zayed Post-Graduate Medical Institute; Sohaib Ashraf, MBBS, Principal Investigator — Shaikh Zayed Post-Graduate Medical Institute
Locations (1):
- Shaikh Zayed Post-Graduate Medical Institute, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No